CLINICAL TRIAL: NCT03611634
Title: Consitution Of A Biological Collection From Samples From The Gut Microbiote In Patients Having A Bone Or Joint Infection Treated By A Suppressive Subcutaneous Antibiotherapy With Betalactamine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, Clinical Research Assistant, Hospices Civils de Lyon
Other Study IDs: 18-126
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Bone and Joint Infection
Keywords: gut microbiote, bone and joint infection, antibiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BIOLOGICAL COLLECTION FROM THE GUT MICROBIOTE: The aim of this study is just to constitute a biological collection from samples from the GUT microbiote in patients having a bone or joint infection treated by a suppressive subcutaneous antibiotherapy with betalactamine. No analysis will be done for instance.
  Interventions: Other: BIOLOGICAL COLLECTION FROM THE GUT MICROBIOTE

INTERVENTIONS:
Other: BIOLOGICAL COLLECTION FROM THE GUT MICROBIOTE — collection of saddles

SUMMARY:
Optimal surgical therapy (debridement in chronic osteomyelitis; device exchange in patients with chronic prosthetic joint infection [PJI]) could be sometimes non-feasible, especially in the elderly population. Therefore, a medical therapy with oral prolonged suppressive antibiotic therapy (PSAT) seems to be an option to prevent recurrence and prosthesis loosening. Unfortunately, some patients are infected with resistant pathogens for which oral antibiotics are not suitable. Subcutaneous (SC) administration of injectable intravenous antibiotics as PSAT could be a convenient way to limit catheter-related complications and facilitate ambulatory care.

However, there are few data concerning the development of resistance under subcutaneous prolonged treatment with betalactamine.

The aim of this study is is just to constitute a biological collection from samples from the GUT microbiote in patients having a bone or joint infection treated by a suppressive subcutaneous antibiotherapy with betalactamine. Later analysis will be led on those samples to detect the acquisition of resistance or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients having an ostéo-articular infection (on material or on native bone) and having an indication of antibiotic treatment suppressive subcutaneous by betalactamine and managed at the Croix-Rousse Hospital
* Patients not opposed to participate to the study

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having a bone or joint infection treated by a suppressive subcutaneous antibiotherapy with betalactamine
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-07-19 (Actual); Primary Completion 2023-07-19 (Estimated); Study Completion 2024-07-19 (Estimated)

PRIMARY OUTCOMES:
BIOLOGICAL COLLECTION FROM SAMPLES FROM THE GUT MICROBIOTE | 36 months
  The aim of this study is just to constitute a biological collection from samples from the GUT microbiote in patients having a bone or joint infection treated by a suppressive subcutaneous antibiotherapy with betalactamine. No analysis will be done for instance.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, Md,PhD, Principal Investigator — Hospices Civils de Lyon - Hopital de la Croix Rousse
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided